CLINICAL TRIAL: NCT00859053
Title: Single-Dose Pharmacokinetics of BMS-790052 in Subjects With Hepatic Impairment Compared to Healthy Subjects
Brief Title: Single-Dose Pharmacokinetics of BMS-790052 in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI444-013
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-790052 in Child-Pugh A (Active Comparator)
  Interventions: Drug: BMS-790052
- BMS-790052 in Child-Pugh B (Active Comparator)
  Interventions: Drug: BMS-790052
- BMS-790052 in Child-Pugh C (Active Comparator)
  Interventions: Drug: BMS-790052
- BMS-790052 in Healthy Subjects (Active Comparator)
  Interventions: Drug: BMS-790052

INTERVENTIONS:
Drug: BMS-790052 — Capsules, Oral, 30 mg, single dose, one day

SUMMARY:
The purpose of this study is to assess the effects of hepatic impairment on the single dose pharmacokinetics of BMS-790052.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects aged 18 to 70 years, with hepatic impairment conforming to Child-Pugh class A, B or C
* Healthy subjects to the extent possible matched to the first four hepatically impaired subject in each Child-Pugh class with regard to age (approximately ± 10 years), body weight (approximately ± 20%) and gender

Key Exclusion Criteria:

* History of esophageal and gastric variceal bleeding within past 6 months
* Primarily cholestatic liver diseases
* Active alcoholic hepatitis
* Stable encephalopathy of >= Stage 2
* Presence of severe ascites or edema
* Presence of hepatopulmonary or hepatorenal syndrome
* Positive for HCV, unless HCV RNA is undetectable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Advanced Clinical Research Institute, Anaheim, California
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 46 participants were enrolled in the study, of which 30 participants were treated with study drug and 16 participants were not treated with study drug as they no longer met study criteria.
Groups:
- Child Pugh Class-A: Participants with mild liver damage were administered with single oral dose of 30 milligrams (mg) (3 x 10 mg capsules) of BMS-790052 after 10 hours overnight fasting.
- Child Pugh Class-B: Participants with moderate liver damage were administered with single oral dose of 30 mg (3 x 10 mg capsules) of BMS-790052 after 10 hours overnight fasting.
- Child Pugh Class-C: Participants with severe liver damage were administered with single oral dose of 30 mg (3 x 10 mg capsules) of BMS-790052 after 10 hours overnight fasting.
- Healthy Participants: Healthy participants were administered with single oral dose of 30 mg (3 x 10 mg capsules) of BMS-790052 after 10 hours overnight fasting.
Period: Overall Study
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Started | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done in safety population, defined as all the participants who received study medication.
Groups:
- Child Pugh Class-A: Participants with mild liver damage were administered with single oral dose of 30 mg (3 x 10 mg capsules) of BMS-790052 after 10 hours overnight fasting.
- Total: Total of all reporting groups
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants | Total
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 30
Age, Customized [Number; unit: participants]
  < 65 years | 6 | 5 | 5 | 12 | 28
  >= 65 years | 0 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 5 | 12
  Male | 4 | 3 | 4 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of BMS-790052
Description: Maximum observed plasma concentration following drug administration from the raw plasma concentration-time data. The plasma samples were analysed for BMS-790052 by using a validated liquid chromatography tandem mass spectrometric (LC-MS/MS) assay.
Time Frame: Pre-dose (0), 0.5,1, 1.5, 2, 4, 8, 12, 24, 48, 72 hours post-dose (both healthy and hepatically impaired participants) and 96 hours post-dose (only for hepatically impaired participants)
Population: Analysis was performed in the Pharmacokinetic population (all participants who received study drug and had adequate PK profiles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
nanograms/milliliter (ng/mL) | 380 (44) | 382 (23) | 317 (65) | 698 (30)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Last Measurable Concentration [AUC(0-T)] of BMS-790052
Description: AUC(0-T) was calculated by the sum of linear trapezoids using non-compartmental analysis.
Time Frame: Pre-dose (0), 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72 hours post-dose (both healthy and hepatically impaired participants) and 96 hours post-dose (only for hepatically impaired participants)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour (h)/mL
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
ng*hour (h)/mL | 4151 (43) | 4490 (38) | 4534 (74) | 7165 (24)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of BMS-790052
Description: AUC(INF) was estimated as AUC(0-T) + Ct/λ z, where λ z was the terminal elimination rate constant and Ct was the last observable concentration.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng* h/mL
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
ng* h/mL | 4174 (43) | 4550 (39) | 4649 (78) | 7286 (25)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of BMS-790052
Description: Tmax was defined as the time required to reach maximum observed plasma concentration. Tmax was directly determined from the raw plasma concentration-time data.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
hours | 1.5 [1 to 2] | 1.0 [1 to 4] | 1.5 [1 to 4] | 1.3 [1 to 2]

5. Primary Outcome: Terminal Half-life (T-HALF) of BMS-790052
Description: Terminal half-life was the time required for one half of the total amount of administered drug eliminated from the body.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
hours | 12.3 (2.49) | 15.0 (4.59) | 17.2 (10.55) | 12.4 (2.23)

6. Primary Outcome: Apparent Total Body Clearance (CLT/F) of BMS-790052
Description: Apparent total body clearance was calculated as dose/AUC(INF). AUC(INF) was estimated as AUC(0-T) + Ct/λ z, where λ z was the terminal elimination rate constant and Ct was the last observable concentration.
Time Frame: as for outcome 1
Population: Analysis was performed in PK set population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/minute (mL/min)
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
milliliter/minute (mL/min) | 120 (85) | 110 (47) | 108 (78) | 69 (29)

7. Primary Outcome: Apparent Clearance of Free BMS-790052 (CLu/F)
Description: CLu/F was calculated by dividing the apparent total body clearance (CLT/F) by mean fraction of unbound drug (fu) for both (1 hour and 4 hour post dose) time points combined. Apparent total body clearance was calculated as dose/AUC(INF). AUC(INF) was estimated as AUC(0-T) + Ct/ λz, where λz was the terminal elimination rate constant and Ct was the last observable concentration.
Time Frame: as for outcome 2
Population: Analysis was performed in PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
mL/min | 19529 (66) | 12028 (52) | 12468 (61) | 11796 (33)

8. Primary Outcome: The Apparent Volume of Distribution at Steady State (Vss/F)
Description: Apparent volume of distribution was calculated by dividing the product of the dose and mean residence time (MRT) by AUC(INF). AUC(INF) was estimated as AUC(0-T) + Ct/λ z, where λ z was the terminal elimination rate constant and Ct was the last observable concentration.
Time Frame: as for outcome 2
Population: Analysis was performed in PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
mL | 98557 (67) | 111612 (24) | 123034 (56) | 61250 (19)

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), and Who Died
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a pre-existing condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Study Discharge (end of study) was Day 4 (healthy participants) or Day 5 (hepatically impaired participants).
Time Frame: Day 1 to end of study for AEs and, Day 1 to up to 30 days after last dose for SAE.
Population: Analysis was done in safety population, defined as all the participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Number analyzed (Participants) | 6 | 6 | 6 | 12
Participants
  SAEs | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Child Pugh Class-A | Child Pugh Class-B | Child Pugh Class-C | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 2/6 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Child Pugh Class-A (N=6) | Child Pugh Class-B (N=6) | Child Pugh Class-C (N=6) | Healthy Participants (N=12)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.